CLINICAL TRIAL: NCT04692402
Title: Feasibility Trial Evaluating Efficacy and Safety of Solitaire™ Thrombus Retrieval Device in the Management of Refractory Thrombus in Patients With Acute Coronary Syndrome
Acronym: Solitaire
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Paul Ong (Other)
Responsible Party: Sponsor-Investigator, Paul Ong, Consultant Cardiologist and Cathlab Director, Tan Tock Seng Hospital
Organization: Tan Tock Seng Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSRB 2018/00865
Record Dates: First submitted 2020-10-28; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Refractory Thrombus in Patients With Acute Coronary Syndrome

STUDY DESIGN:
Masking Description: Investigator initiated multicentre open label prospective feasibility trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- open label (Other): open label prospective feasibility trial.
  Interventions: Device: Solitaire™ thrombus retrieval device

INTERVENTIONS:
Device: Solitaire™ thrombus retrieval device — After consent has been obtained, interventional cardiologist selects the proper solitaire device size per device-specific instructions for use. Adjunctive intervention with Solitaire will be done with a maximum of 2 device deployments. Do not perform more than three recovery attempts in the same vessel using the devices (Maximum of 2 attempts per device per subject). Do not reposition each device more than two times. TIMI flow, thrombus grade and myocardial blush grade will be assessed immediately upon completion of procedure. If recanalization is deemed inadequate by the interventional cardiologist, rescue treatment will follow as per current clinical practice. All other procedures followed will be as clinically indicated.

SUMMARY:
The study is designed as a multicentre open label prospective feasibility trial to capture preliminary efficacy and safety information on Solitaire device to plan an appropriate pivotal study.

DETAILED DESCRIPTION:
We hypothesize that Solitaire device could be effectively and safely used as an adjunctive interventional technique in ACS patients found to have refractory thrombus during PCI.

1. Primary Objectives To evaluate intra-procedure efficacy of using Solitaire in ACS patients with refractory thrombus.
2. Secondary Objectives To evaluate clinical efficacy of using Solitaire in ACS patients with refractory thrombus, up to one year post-procedure.

To evaluate safety of using Solitaire in ACS patients with refractory thrombus.

The target enrolment is 51 patients diagnosed with STEMI, NSTEMI or UA and found to have refractory thrombus during PCI. Eligible patients will be identified at the ED or Inpatient ward of the 5 participating hospitals. The projected enrolment period is for two years and follow up for one year. A screening log will be maintained at each site to keep record of patients who were eligible for the study but not enrolled, to establish any selection bias.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the inclusion criteria listed below will be included in this study:

1. Index event of ST segment elevation or non-ST segment elevation MI or Unstable Angina defined as:

   1. Presentation to hospital with symptoms of myocardial ischemia (Chest pain or angina equivalent) lasting for ≥10 minutes at rest

      AND 1 of the following:
   2. Persistent ST segment elevation ≥1mm (0.1 mV) in two or more contiguous limb leads or ≥2mm (0.2 mV) in ) in one or more contiguous precordial leads OR
   3. New or presumed new left bundle branch block (LBBB) OR
   4. ST segment depression ≥1mm (0.1 mV) in two or more contiguous leads (not known to be pre-existing or due to a known cause such as LV hypertrophy or digoxin) OR
   5. Troponin T or I greater than the laboratory upper normal limit.
2. Referred for urgent or emergency PCI AND Thrombus burden of TG 4 or above OR TIMI flow grade of 1 or less in at least one native infarct related artery following either

   1. Manual aspiration thrombectomy OR
   2. Balloon Angioplasty OR
   3. AngioJet RT OR
   4. Patient having deferred PCI due to heavy thrombus but continue to demonstrate recalcitrant thrombus upon repeat angiography.

Exclusion Criteria:

Subjects meeting any of the exclusion criteria listed below will be excluded from this study:

1. Age ≤ 21 years
2. Cardiogenic shock
3. killip class 3 or above at presentation
4. Known relative contraindications for the use of Solitaire:

   1. Prior stent in infarct related artery
   2. Significant proximal stenosis OR Ostial lesion at angiography
   3. Extensive calcification
5. Life expectancy less than six months due to non-cardiac condition
6. Participants categorised as vulnerable subjects (ex: prisoners, pregnant women, and mentally disabled persons)
7. Patients at high risk of being lost to follow up (ex: non-residents)
8. Participation in any study with an investigational drug or device within the last 30 days
9. Patients who are unable to provide informed consent prior to any procedure .

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2019-07-16 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of successful recanalization defined as an immediate post-procedure Thrombolysis in Myocardial Infarction (TIMI) flow of 2 or 3. | immediate post-procedure
  Primary Efficacy Endpoint
Occurrence of any stroke | immediate post-procedure up to 30 days
  Occurrence of any stroke, defined as the presence of a new focal neurologic deficit thought to be vascular in origin, with signs or symptoms lasting more than 24 hours, from immediate post-procedure up to 30 days.
Incidence of study device-related Serious Adverse Events (SAEs) up to 30 days. | up to 30 days
  Primary Safety Endpoint
Incidence of emboli in new territory (ENT) at 24 hrs ± 8 hrs post procedure (ENT: Embolization territories outside of the target downstream territory). | at 24 hours ± 8 hours post procedure
  Primary Safety Endpoint

SECONDARY OUTCOMES:
Rate of successful thrombus resolution defined as an immediate post-procedure thrombus burden of thrombus grade (TG) 1 or less | immediate post-procedure
  Secondary Endpoints
Rate of successful recanalization defined as a reduction in corrected TIMI frame count after use of the Solitaire device. | immediate post-procedure
  Secondary Endpoints
Rate of successful myocardial perfusion defined as an immediate post-procedure myocardial blush grade (MBG) of 2 or more | immediate post-procedure
  Secondary Endpoints
Rate of device success defined as successful delivery and retrieval of the device without complication | immediate post- procedure
  Secondary Endpoints
Occurrence of major adverse cardiac and cerebrovascular events (MACCE) | up to one year post-procedure
  Occurrence of major adverse cardiac and cerebrovascular events (MACCE), defined as composite of all cause death, myocardial infarction, target vessel revascularisation or stroke, up to one year post-procedure.
All-cause mortality through 90 days post procedure. | 90 days post procedure
  Secondary Endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Paul Jau Lueng Ong, Principal Investigator — Paul Ong Jau Lueng
Locations (5):
- Singapore (5):
  - National Heart Centre Singapore (NHCS), Singapore, Singaproe
  - National University Heart Centre Singapore (NUHCS), Singapore
  - Tan Tock Seng Hospital (TTSH), Singapore
  - Changi General Hospital (CGH) Changi General Hospital, Singapore
  - Khoo Teck Puat Hospital, Singapore